CLINICAL TRIAL: NCT01999530
Title: Exploring the Effects of Prazosin on Basal Dopamine in Healthy Humans: A [11C]-(+)-PHNO PET Pilot Study
Brief Title: The Effects of Prazosin on Dopamine in Healthy Humans: A PET Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Lung Association (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Bernard Le Foll, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 224/2012
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Healthy
Keywords: prazosin; dopamine; healthy; Positron Emission Tomography; PHNO; scan; effect
MeSH Terms: interventions — Prazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prazosin Hydrochloride (Experimental): Gradual upward titration to 15mg/day (or highest dose tolerated) for approximately three weeks.
  Interventions: Drug: Prazosin Hydrochloride

INTERVENTIONS:
Drug: Prazosin Hydrochloride — Gradual upward titration to 15mg/day for approximately three weeks.
  Other Names: Teva-Prazosin; Prazosin; Minipress

SUMMARY:
The purpose of this study is to find out whether short term treatment with a antihypertensive medication prazosin, can influence the levels of a dopamine in the brain. We will examine the levels of dopamine in the the brain using Positron Emission Tomography (PET) and Magnetic Resonance Imaging (MRI). We hypothesize that there will be no significant changes in dopamine levels in healthy individuals taking prazosin.

DETAILED DESCRIPTION:
The purpose of this study is to find out whether short term treatment with a antihypertensive medication prazosin, can influence the levels of dopamine in the brain. We will examine the levels of dopamine in the the brain using Positron Emission Tomography (PET) and Magnetic Resonance Imaging (MRI). The study will involve three PET scans and one MRI. One PET scan will be performed before the participants take prazosin for approximately three weeks, and the last two PET scans will be performed after the prazosin medication phase. We hypothesize that there will be no significant changes in dopamine levels in healthy individuals taking prazosin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females of any ethnic origin between 19 and 45 years old

Exclusion Criteria:

* Use of any illicit drugs in past 3 months prior to randomization and/or have a current or past diagnosis of drug abuse/dependence (including alcohol)
* Current or past DSM-IV diagnosis of any Axis I psychiatric disorder
* Major psychiatric illness and/or substance dependence in first order relatives
* Current active or past suicidal ideation
* Baseline systolic blood pressure outside the normal range
* Current use of medications that could interact with prazosin (e.g. beta blockers, phosphodiesterasetype 5 inhibitors, indomethacin, verapamil, modafinil, clonidine)
* Current use or use during the previous month of medication that may affect the CNS at the time of scanning (e.g. neuroleptics, bupropion)
* Any significant abnormalities in baseline blood results (e.g. CBC, renal and hepatic indicators) or ECG readings that would preclude the use of prazosin
* Pregnancy, trying to become pregnant or breastfeeding
* Presence of metal objects in the body (e.g. some artificial joints, bone pins, surgical clips, skull plate, certain part of dental braces) or implanted electronic devices (e.g. cardiac pacemaker, neurostimulator), that preclude safe MR scanning
* Claustrophobia
* Participation in any nuclear medicine procedures that, including the dose received during participation in this study, will bring the total radiation dose over the currently approved guideline of 20mSv in a 12-month period
* Cardiovascular or cerebrovascular diseases
* History of or current neurological illnesses including seizure disorders, migraine, multiple sclerosis, movement disorders, head trauma, CVA or CNS tumor
* Abnormal body mass (defined as not within 20% of normal BMI
* Learning disability, amnesia or other conditions that impede memory and attention

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching — http://www.camh.net/research
- Available data/document: Publication — https://www.ncbi.nlm.nih.gov/pubmed/28233334

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prazosin Hydrochloride
Started | 20
Completed | 7
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Prazosin Hydrochloride
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1
  Caucasian | 3
  Hispanic | 2
  Mixed | 1
Region of Enrollment [Number; unit: participants]
  Canada | 7

OUTCOME MEASURES:

1. Primary Outcome: Changes in [11C]-(+)-PHNO Binding (Measured as Binding Potential) in Dorsal Caudate (DC)
Description: Binding potential (an estimate of the ratio of Bmax/kd) was measured by positron emission tomography to determine if taking prazosin alters the amount of tracer bound to receptors. A negative change in binding potential means a decrease in binding potential and a positive change in binding potential represents an increase. Bmax is the total density of receptors. kd is the affinity of a drug for the target
Time Frame: 3 weeks after taking prazosin
Measure: Mean (Full Range); unit: binding potential
Arm/Group | Prazosin Hydrochloride
Number analyzed (Participants) | 7
binding potential | 2.1 [1.4 to 2.8]

ADVERSE EVENTS:
Arm/Group | Prazosin Hydrochloride
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 6/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prazosin Hydrochloride (N=20)
Nausea (Gastrointestinal disorders) | 6 — Adverse events caused by prazosin

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No